CLINICAL TRIAL: NCT02554981
Title: Evaluation of Maintaining Visual Performance Of Subjects Who Engage in Electronic Visual Tasking While Using Restasis (EMPOWER)
Brief Title: Evaluation of Maintaining Visual Performance in Participants Who Engage in Electronic Visual Tasking While Using Restasis®
Acronym: EMPOWER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-RES-015-001
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RESTASIS® (Experimental): 1 drop of RESTASIS® ophthalmic emulsion instilled in each eye twice a day for 6 months.
  Interventions: Drug: Cyclosporine 0.05% Ophthalmic Emulsion

INTERVENTIONS:
Drug: Cyclosporine 0.05% Ophthalmic Emulsion — Cyclosporine 0.05% Ophthalmic Emulsion (RESTASIS®) 1 drop instilled in each eye twice a day.
  Other Names: RESTASIS®

SUMMARY:
This study will evaluate the efficacy of Restasis® in participants with dry eye disease who engage in electronic visual tasking.

ELIGIBILITY:
Inclusion:

* Has Eye Symptoms when using video display terminals
* Has a reported history of dry eye in both eyes.

Exclusion:

* Diagnosed with eye infection or active inflammation.
* Has worn contact lenses within the past 7 days or anticipated use during the study.
* Has used any eye drops within 2 hours.
* Has had laser-assisted in situ keratomileusis (LASIK) within 12 months.
* Has used Restasis® within 90 days.
* Has had any eye and or/lid surgeries within 6 months.
* Has had cataract surgery in either eye.
* Has current punctal occlusion or anticipate a change in punctal occlusion status at any point during the study.
* Is currently taking any topical ophthalmic prescriptions or over-the-counter solutions, artificial tears, gels or lid scrubs that cannot be discontinued for the trial duration.
* Use of medication known to cause ocular drying that is not on a stable dose for at least 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2016-03-24 (Actual); Study Completion 2016-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jai Parekh, Study Director — Allergan
Locations (2):
- United States (2):
  - Andover Eye Associates, Inc, Andover, Massachusetts
  - Total Eye Care, PA, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RESTASIS®
Started | 51
Completed | 46
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Administrative Reasons | 1
Not completed — Other Miscellaneous Reasons | 3

BASELINE CHARACTERISTICS:
Population: 51 participants were initially enrolled in the study, 1 participant discontinued before dosing and is not included in the Intent-to-treat (ITT) population.
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Corneal Staining Score With Fluorescein in the Worse Eye
Description: Total corneal staining with fluorescein was measured in the worse eye using the Ora Calibra™ (Scale 1.0) 5-point scale where 0= none (best), no staining to 4=severe staining (worst). The sum of the total includes 3 regions of the cornea, resulting in a maximum possible score of 12 (severe staining score of 4 in all three regions). The worse eye is defined as the worst eye at Baseline. A negative change from Baseline represents a decrease in staining (improvement).
Time Frame: Baseline, Month 6
Population: ITT population included all enrolled participants who received at least one dose of the study drug. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
score on a scale
  Baseline | 7.05 (1.011)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | -1.51 (1.466)

2. Primary Outcome: Change From Baseline in the Total Conjunctival Staining Score With Fluorescein in the Worse Eye
Description: Total conjunctival staining with fluorescein was measured in the worse eye using the Ora Calibra™ (Scale 1.0) 5-point scale where 0= none (best), no staining to 4=severe staining (worst). The sum of the total includes 2 regions of the conjunctiva, resulting in a maximum possible score of 8 (severe staining score of 4 in both regions). The worse eye is defined as the worst eye at Baseline. A negative change from Baseline represents a decrease in staining (improvement).
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
score on a scale
  Baseline | 4.57 (1.237)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | -0.61 (1.238)

3. Primary Outcome: Change From Baseline in the Central Region Staining Score With Fluorescein in the Worse Eye
Description: Staining with fluorescein in the central region of the eye was measured in the worse eye using the Ora Calibra™ (Scale 1.0) 5-point scale where 0= none (best), no staining to 4=severe staining (worst). The worse eye is defined as the worst eye at Baseline. A negative change from Baseline represents a decrease in staining (improvement).
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
score on a scale
  Baseline | 2.29 (0.441)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | -0.75 (0.656)

4. Primary Outcome: Change From Baseline in the Total Corneal Staining Score With Lissamine Green in the Worse Eye
Description: Total corneal staining with lissamine green was measured in the worse eye using the Ora Calibra™ (Scale 1.0) 5-point scale where 0= none (best), no staining to 4=severe staining (worst). The sum of the total includes 3 regions of the cornea, resulting in a maximum possible score of 12 (severe staining score of 4 in all three regions). The worse eye is defined as the worst eye at Baseline. A negative change from Baseline represents a decrease in staining (improvement).
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
score on a scale
  Baseline | 4.00 (1.378)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | -0.34 (1.418)

5. Primary Outcome: Change From Baseline in the Total Conjunctival Staining Score With Lissamine Green in the Worse Eye
Description: Total conjunctival staining with lissamine green was measured in the worse eye using the Ora Calibra™ (Scale 1.0) 5-point scale where 0= none (best), no staining to 4=severe staining (worst). The sum of the total includes 2 regions of the conjunctiva, resulting in a maximum possible score of 8 (severe staining score of 4 in both regions). The worse eye is defined as the worst eye at Baseline. A negative change from Baseline represents a decrease in staining (improvement).
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
score on a scale
  Baseline | 3.99 (1.486)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | -0.18 (1.235)

6. Primary Outcome: Change From Baseline in the Central Region Staining Score With Lissamine Green in the Worse Eye
Description: Staining with lissamine green in the central region of the eye was measured in the worse eye using the Ora Calibra™ (Scale 1.0) 5-point scale where 0= none (best), no staining to 4=severe staining (worst). The worse eye is defined as the worst eye at Baseline. A negative change from Baseline represents a decrease in staining (improvement).
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
score on a scale
  Baseline | 0.85 (0.822)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | -0.24 (0.524)

7. Primary Outcome: Change From Baseline in Font Size
Description: The minimum font (letter) size read correctly was assessed. Smaller font size (less points) indicates better ability. A negative change from Baseline indicates an improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline, Month 6
Population: ITT population was defined as all enrolled participants who received at least one dose of study drug. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
points
  Baseline | 9.0 (0.00)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | 0.0 (0.21)

8. Primary Outcome: Change From Baseline in Words Read Incorrectly
Description: The numbers of words read incorrectly are counted. A positive change from Baseline indicates a worsening (more words read incorrectly) and a negative change from Baseline indicates an improvement.
Time Frame: Baseline, Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: incorrect words
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
incorrect words
  Baseline | 16.6 (22.00)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | -4.1 (16.64)

9. Primary Outcome: Change From Baseline in Time to Read Passage
Description: The time to read passage (selected portion of text ) in seconds was assessed. A negative change from Baseline indicates an improvement (less time to read the passage).
Time Frame: Baseline, Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
seconds
  Baseline | 126.0 (28.64)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | -0.7 (24.48)

10. Primary Outcome: Change From Baseline in Reading Rate
Description: Reading speed was assessed as the number of words read correctly calculated as words/minute. A positive change from Baseline indicates an improvement (more words read correctly/minute) and a negative change from Baseline indicates a worsening (less words read correctly/minute).
Time Frame: Baseline, Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: correct words/minute
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
correct words/minute
  Baseline | 146.6 (64.18)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | -3.6 (69.80)

11. Secondary Outcome: Change From Baseline in Tear Film Break Up Time (TFBUT) in the Worse Eye
Description: TFBUT is defined as the time required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film. The worse eye is defined as the Worse Eye at Baseline. A positive number change from Baseline indicates improvement and a negative number change from Baseline indicates a worsening.
Time Frame: Baseline, Month 6
Population: ITT population included all enrolled participants who received at least one dose of study drug. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
seconds
  Baseline | 2.38 (1.073)
  Change from Baseline at Month 6: number analyzed (Participants) | 46
  Change from Baseline at Month 6 | -0.31 (1.258)

12. Secondary Outcome: Change From Baseline in Ocular Protection Index (OPI) 2.0 in the Worse Eye
Description: A device was used to assess OPI 2.0. This technology measures blink and tear film break-up area. These values demonstrate the average area of tear deficiency/corneal exposure. The worse eye is defined as the worse eye at Baseline. A negative value indicates an improvement in corneal protection.
Time Frame: Baseline, Month 6
Population: Participants from the ITT population, all enrolled participants who received at least one dose of study drug with data available for analysis. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: percent of area
Arm/Group | RESTASIS®
Number analyzed (Participants) | 49
percent of area
  Baseline | 1.38 (2.064)
  Change from Baseline at Month 6: number analyzed (Participants) | 40
  Change from Baseline at Month 6 | -0.87 (1.975)

13. Secondary Outcome: Change From Baseline in Interblink Interval (IBI) in the Worst Eye
Description: A device was used to assess IBI. The IBI measures the time in seconds between blinks in the worse eye. A positive number change from baseline indicates a worsening (more frequent blinks) and a negative number change from baseline (less frequent blinks) indicates an improvement.
Time Frame: Baseline, Month 6
Population: ITT population included all enrolled participants who received at least 1 dose of study drug. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RESTASIS®
Number analyzed (Participants) | 49
seconds
  Baseline | 5.27 (6.052)
  Change from Baseline at Month 6: number analyzed (Participants) | 41
  Change from Baseline at Month 6 | -1.16 (6.399)

14. Secondary Outcome: Change From Baseline in OSDI© Total Score
Description: The OSDI© questionnaire consists of 12 questions measuring the presence of ocular symptoms. Each of the 12 questions was assessed using a 5-point scale (where 0=none of the time and 4=all of the time). The score is converted to a 0 to 100 point score where 0 is no symptoms and 100 is most symptoms. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Month 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
score on a scale
  Baseline | 45.1 (17.76)
  Change from Baseline at Month 6 | -14.9 (16.50)

15. Secondary Outcome: Change From Baseline in Driving at Night on the OSDI©
Description: The OSDI© consists of 12 questions measuring the presence of ocular symptoms. The Driving at Night question was assessed using a 5-point scale (0=none of the time to 4=all of the time). Higher OSDI© scores are associated with greater severity. A negative number change from Baseline indicates improvement and a positive number change from Baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 43
score on a scale
  Baseline | 1.7 (1.30)
  Change from Baseline at Month 6: number analyzed (Participants) | 39
  Change from Baseline at Month 6 | -0.5 (1.14)

16. Secondary Outcome: Change From Baseline in Working With a Computer or Bank Machine on the OSDI©
Description: The OSDI© consists of 12 questions measuring the presence of ocular symptoms. The Working with a Computer or Bank Machine question was assessed using a 5-point scale (0=none of the time to 4=all of the time). Higher OSDI© scores are associated with greater severity. A negative number change from Baseline indicates improvement and a positive number change from Baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 49
score on a scale
  Baseline | 1.9 (1.03)
  Change from Baseline at Month 6: number analyzed (Participants) | 44
  Change from Baseline at Month 6 | -0.8 (1.08)

17. Secondary Outcome: Change From Baseline in Watching Television (TV) on the OSDI©
Description: The OSDI© consists of 12 questions measuring the presence of ocular symptoms. The Watching TV question was assessed using a 5-point scale (0=none of the time to 4=all of the time). Higher OSDI© scores are associated with greater severity. A negative number change from Baseline indicates improvement and a positive number change from Baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 48
score on a scale
  Baseline | 1.8 (1.11)
  Change from Baseline at Month 6: number analyzed (Participants) | 42
  Change from Baseline at Month 6 | -0.9 (1.12)

18. Secondary Outcome: Change From Baseline in Blurred Vision on the OSDI©
Description: The OSDI© consists of 12 questions measuring the presence of ocular symptoms. The Blurred Vision question was assessed using a 5-point scale (0=none of the time to 4=all of the time). Higher OSDI© scores are associated with greater severity. A negative number change from Baseline indicates improvement and a positive number change from Baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
score on a scale
  Baseline | 1.7 (1.18)
  Change from Baseline at Month 6: number analyzed (Participants) | 45
  Change from Baseline at Month 6 | -0.6 (0.86)

19. Secondary Outcome: Change From Baseline in Poor Vision on the OSDI©
Description: The OSDI© consists of 12 questions measuring the presence of ocular symptoms. The Poor Vision question was assessed using a 5-point scale (0=none of the time to 4=all of the time). Higher OSDI© scores are associated with greater severity. A negative number change from Baseline indicates improvement and a positive number change from Baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
score on a scale
  Baseline | 1.5 (1.23)
  Change from Baseline at Month 6: number analyzed (Participants) | 45
  Change from Baseline at Month 6 | -0.5 (0.84)

20. Secondary Outcome: Change From Baseline in Reading on the OSDI©
Description: The OSDI© consists of 12 questions measuring the presence of ocular symptoms. The Reading question was assessed using a 5-point scale (0=none of the time to 4=all of the time). Higher OSDI© scores are associated with greater severity. A negative number change from Baseline indicates improvement and a positive number change from Baseline indicates worsening.
Time Frame: Baseline, Month 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 50
score on a scale
  Baseline | 1.5 (1.25)
  Change from Baseline at Month 6: number analyzed (Participants) | 45
  Change from Baseline at Month 6 | -0.3 (1.15)

21. Secondary Outcome: Change From Baseline in the Ocular Discomfort Scale Post Wilkins Test in the Worst Eye
Description: Participants assessed ocular discomfort post Wilkins Rate of Reading Test using the Ora Calibra™ 5-point scale where 0=no discomfort to 4=constant discomfort. A positive number change from Baseline indicates a worsening and a negative number change from Baseline indicates an improvement.
Time Frame: Baseline, Month 6
Population: Participant from the ITT population, all enrolled participants who received at least one dose of study drug, with data available for analysis. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESTASIS®
Number analyzed (Participants) | 49
score on a scale
  Baseline | 3.08 (1.017)
  Change from Baseline at Month 6: number analyzed (Participants) | 45
  Change from Baseline at Month 6 | -0.60 (1.232)

ADVERSE EVENTS:
Arm/Group | RESTASIS®
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 6/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RESTASIS® (N=50)
Papillary thyroid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Peripheral vascular disease (Vascular disorders) | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RESTASIS® (N=50)
Visual acuity reduced (Eye disorders) | 3
Nasopharyngitis (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.